CLINICAL TRIAL: NCT01813110
Title: Effects of a Prescription Omega-3 Fatty Acid Concentrate in a Placebo-controlled Trial of Human Endotoxemia
Brief Title: Effects of a Prescription Omega-3 Fatty Acid Concentrate on Induced Inflammation
Acronym: PRONOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PRONOVA
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Inflammatory Responses
Keywords: inflammation; omega-3; fish oil
MeSH Terms: conditions — Inflammation | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Identical olive oil capsules
  Interventions: Drug: Placebo
- Omega-3 (Experimental): 4 g prescription omega-3 concentrate (4 g/d prescription omega-3 fatty acid concentrate taken orally for 8-12 weeks)
  Interventions: Drug: 4 g prescription omega-3 concentrate

INTERVENTIONS:
Drug: 4 g prescription omega-3 concentrate — 4 g/d prescription omega-3 fatty acid concentrate taken orally for 8-12 weeks
  Other Names: Lovaza; Omacor
  Arms: Omega-3
Drug: Placebo — olive oil
  Other Names: No other name (control)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether the marine omega-3 fatty acids can attenuate inflammatory responses to endotoxin challenge.

DETAILED DESCRIPTION:
Controlled endotoxin infusion has been used widely as a model system to evaluate anti-inflammatory mediators and therapies in a controlled, in vivo setting. It is well established that infusion of bacterial endotoxin (also known as lipopolysaccharide or LPS) in humans results in a marked increase in inflammatory cytokines, most notably TNF-α, IL-1, IL-6 and IL-8, CRP, granulocyte colony stimulating factor (GCSF); eicosanoids, such as prostaglandin (PG) E2 and other mediators. Administration of endotoxin, even at a low dose (0.6 ng/kg) elevates circulating concentrations of inflammatory cytokines, and mimics the inflammatory effects of chronic diseases. This model has been used for decades and has proved to be safe and informative for evaluating anti-inflammatory therapeutic interventions on human inflammation and downstream consequences.

Prolonged or chronic inflammation is involved in the etiology of several diseases such as cardiovascular disease (CVD), diabetes, rheumatoid arthritis, cancer, and neurodegenerative diseases such as Alzheimer's disease. The evidence base clearly demonstrates benefits of diet in ameliorating inflammation and reducing the burden of chronic disease. With respect to marine-derived omega-3 fatty acids and various markers of inflammation related to cardiovascular disease (CVD), both population studies and randomized controlled supplementation trials have yielded mixed results. It is well established that these omega-3 fatty acids are precursors of series-3 prostanoids, thromboxanes, 5-series leukotrienes, and novel lipid mediators such as resolvins and protectins that have anti-inflammatory effects. We hypothesize that supplementation of omega-3 fatty acids will blunt the response to an inflammatory stimulus and/or enhance the resolution phase.

We propose to test this hypothesis using an in vivo endotoxin challenge with a pharmacological dose of omega-3 fatty acid ethyl esters (P-OM3, 3.4 g/d EPA + DHA) in healthy volunteers. Our proposed approach is novel in that we will provoke an in vivo inflammatory response by infusing human subjects with a low dose (0.6 ng/kg body weight) of sterile endotoxin (lipopolysaccharide [LPS]) in contrast to studies that have attempted to reverse established inflammatory pathology. Results from our proposed research will advance our understanding of the effect of omega-3 fatty acids on prevention/attenuation of an inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Men between the ages of 20 and 45.
2. BMI ≥20 and ≤30
3. Participants who are able to give written informed consent and willing to comply with all study-related procedures.
4. Any race or ethnic background is acceptable
5. Non-smoking

The specific exclusion criteria are:

1. Previous history of vasovagal reactions or unprovoked fainting (I.e. fainting as a result of prolonged standing, exercise)
2. Resting heart rate < 55 bpm
3. History of atherosclerotic cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease
4. History of diabetes mellitus (and/or a fasting glucose >126 mg/dL at screening)
5. Chronic anti-inflammatory medication use or treatment with aspirin, NSAIDs, COX-2 inhibitors; steroids or any immunomodulatory therapy 2 weeks prior to the screening visit
6. Self-reported history of allergy to fish
7. History of a non-skin malignancy within the previous 5 years
8. Renal insufficiency as defined by creatinine outside of lab defined normal range at Screening Visit
9. History of liver disease or abnormal LFTs (AST, ALT, Alk. Phos., GGT > 1.5x ULN; bilirubin > 2x ULN) at Screening Visit
10. Total white blood cell count less than or equal to 3.0 THO/uL
11. Hemoglobin less than 11.0 g/dL
12. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition or minor active infection
13. Self-reported history of HIV positive
14. Participants who have undergone any organ transplant
15. Individuals who currently use tobacco products or have done so in the previous 30 days.
16. Participants who are unwilling to discontinue use of nutritional supplements, herbs or vitamins unless approved by study staff.
17. Participants who are unwilling to eliminate omega-3 fatty acid (EPA + DHA) supplements and/or fortified food, or have a usual intake of high omega-3 fish (tuna and other non-fried fish) > 2 servings per week
18. Elevated blood pressure (BP > 159/99) or use of any anti-hypertensive medications.
19. Latex allergy
20. Unwillingness to refrain from blood donation for 2 months prior to and following endotoxin administration
21. Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator
22. Inability to take study capsules
23. History of severe, repeated headaches
24. History of migraine
25. Medical condition that causes severe nausea or vomiting
26. Low resting blood pressure (SBP < 90 mmHg)
27. History of atrial fibrillation/flutter
28. Abnormal coagulation parameters (platelet count, prothrombin time with INR), documented coagulation abnormality, or use of anticoagulant medication
29. High LDL-C (> or = 160 mg/dL)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jensen, MD, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A balanced randomization scheme was developed in advance, and subjects were assigned to a treatment sequence at enrollment.
Groups:
- Placebo (8 Weeks), Then Omega-3 Fatty Acids (8 Weeks): 8 weeks of placebo (olive oil) supplementation followed by 8 weeks of omega-3 fatty acid supplementation (4 g prescription omega-3 fatty acid concentrate)
- Omega-3 Fatty Acids (8 Weeks), Then Placebo (8 Weeks): 8 weeks of omega-3 fatty acid supplementation (4 g prescription omega-3 fatty acid concentrate) followed by 8 weeks of placebo (olive oil) supplementation
Period: Overall Study
Arm/Group | Placebo (8 Weeks), Then Omega-3 Fatty Acids (8 Weeks) | Omega-3 Fatty Acids (8 Weeks), Then Placebo (8 Weeks)
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only the 20 participants who completed the study are included in the baseline characteristics analysis
Groups:
- Baseline: Baseline (prior to placebo or omega-3 supplementation)
Arm/Group | Baseline
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in C Reactive Protein (CRP)
Description: Change in blood levels of CRP at 24 hours post endotoxin administration, after each 8 week intervention
Time Frame: 24 hours post endotoxin administration, following each 8 week intervention
Measure: Mean (Standard Error); unit: mg/L
Groups:
- Placebo (8 Weeks): 8 weeks of placebo (olive oil) supplementation prior to low-dose endotoxin challenge
- Omega-3 Fatty Acids (8 Weeks): 8 weeks of omega-3 fatty acid supplementation (4 g prescription omega-3 fatty acid concentrate) prior to low-dose endotoxin challenge
Arm/Group | Placebo (8 Weeks) | Omega-3 Fatty Acids (8 Weeks)
Number analyzed (Participants) | 20 | 20
mg/L | 17.2 (1.8) | 17.1 (1.8)

2. Secondary Outcome: Tumor Necrosis Factor-α (TNF-α)
Description: Change in the plasma concentration of TNF-α at 2 hours post endotoxin administration, after each 8 week intervention
Time Frame: 2 hours post endotoxin administration, following each 8 week intervention
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo (8 Weeks) | Omega-3 Fatty Acids (8 Weeks)
Number analyzed (Participants) | 20 | 20
pg/mL | 58.3 (8.1) | 59.9 (8.1)

3. Secondary Outcome: Interleukin-6 (IL-6)
Description: Change in the plasma concentration of TNF-α at 2 hours post endotoxin administration, after each 8 week intervention
Time Frame: 2 hours post endotoxin administration, following each 8 week intervention
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo (8 Weeks) | Omega-3 Fatty Acids (8 Weeks)
Number analyzed (Participants) | 20 | 20
pg/mL | 90.6 (14.0) | 99.9 (14.0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 1 year.
Description: Adverse event collection was done continuously throughout the study. Participants were seen for a baseline visit and a midpoint visit (~4 weeks into the 8 week intervention period), and for the endotoxin challenge testing they were seen on the day of the injection, and 1, 2, 3, and 7 days post endotoxin administration. Participants were asked to report any adverse events at these visits and were asked to contact study personnel at any time between these specified visits to report any problems.
Groups:
- Placebo, Omega-3: 8 weeks of placebo (olive oil) supplementation followed by 8 weeks of omega-3 fatty acid supplementation (4 g prescription omega-3 fatty acid concentrate
- Omega-3, Placebo: 8 weeks of omega-3 fatty acid supplementation (4 g prescription omega-3 fatty acid concentrate) followed by 8 weeks of placebo (olive oil) supplementation
Arm/Group | Placebo, Omega-3 | Omega-3, Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No